CLINICAL TRIAL: NCT02682134
Title: Comparison Between Xylocaine Gel as Endotracheal Cuff Lubricant Versus Dexamethasone 8 mg Intravenously or Both for Sore Throat Prevention Following Intubation: Interventional Study
Brief Title: Sore Throat Prevention Following Intubation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Aboud Nayef AlJabari, Regional and Cardio-thoracic anesthesia doctor, University of Jordan
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: AAlJabari
Record Dates: First submitted 2016-02-05; First posted 2016-02-15 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Sore Throat
Keywords: Sore Throat; Intubation; Xylocaine; Dexamethasone
MeSH Terms: conditions — Pharyngitis | interventions — Lidocaine; Dexamethasone; Fumigant 93

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Xylocaine "X" (Experimental): Patients received xylocaine gel as lubricant on endotracheal tube
  Interventions: Drug: xylocaine
- Dexamethasone "D" (Experimental): Patients were given dexamethasone 8 mg intravenously
  Interventions: Drug: Dexamethasone
- xylocaine and dexamethasone "XD" (Experimental): Patients were given both xylocaine gel and dexamethasone 8 mg intravenously
  Interventions: Drug: Xylocaine and Dexamethasone

INTERVENTIONS:
Drug: xylocaine — First group were given xylocaine
  Other Names: X
  Arms: Xylocaine "X"
Drug: Dexamethasone — Second group were given Dexamethasone
  Other Names: D
  Arms: Dexamethasone "D"
Drug: Xylocaine and Dexamethasone — Third group were given both Xylocaine and Dexamethasone
  Other Names: XD
  Arms: xylocaine and dexamethasone "XD"

SUMMARY:
The aim of this interventional study is to find out the incidence of sore throat among intubated patients in Jordan university hospital and to find out which is preventive and effective method to decrease sore throat;is it xylocaine gel on endotracheal cuff as lubricant versus dexamethasone 8 mg intravenously or both.

DETAILED DESCRIPTION:
Three groups were divided into: first group received xylocaine gel as endotracheal cuff lubricant,second group received dexamethasone 8 mg intravenously and third group received both( xylocaine and dexamethasone).

The investigator compared between the three groups regarding sore throat in intubated patients and followed them up to 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3.
* Elective VS Emergency.
* Cuffed endo-tracheal tubes.
* Different types of surgery.

Exclusion Criteria:

* Pregnant ladies.
* ICU patients.
* <15 years of age
* Laryngeal mask airway

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Comparison in preventing sore throat: xylocaine gel versus dexamethasone or both following intubation. | 4 months
  Questionnaire follow up in intubated patients.

SECONDARY OUTCOMES:
Sore throat SCALE | 4 months
  Sore throat scale from None,mild,moderate till severe.

CONTACTS AND LOCATIONS:
Overall Officials: Aboud Aljabari, Principal Investigator — University of Jordan

IPD SHARING:
Plan to Share IPD: Yes